CLINICAL TRIAL: NCT03443024
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Evaluate the Efficacy and Safety of Lebrikizumab in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Lebrikizumab (LY3650150) in Participants With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17826; J2T-DM-KGAF (Other: Eli Lilly and Company); DRM06-AD01 (Other: Dermira, Inc)
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 125 milligrams (mg) Lebrikizumab - Every 4 Weeks (Q4W) (Experimental): 125 mg Lebrikizumab administered subcutaneously (SC) once Q4W.
  Baseline: Loading dose 250 mg Lebrikizumab SC (two injections SC 1-milliliter (mL) of 125 mg/mL Lebrikizumab and 1-mL placebo).
  Week 2: Four 1-mL SC injections placebo.
  Weeks 4, 8, 12: 125 mg SC Lebrikizumab and 1-mL SC placebo.
  Weeks 6, 10, 14: Two 1-mL SC placebo.
  Interventions: Biological: Lebrikizumab; Drug: Placebo
- 250 mg Lebrikizumab - Q4W (Experimental): 250 mg Lebrikizumab administered SC once Q4W.
  Baseline: Loading dose of 500 mg (four 1-mL SC injections of 125 mg/mL Lebrikizumab).
  Week 2: Four 1-mL SC injections of placebo.
  Weeks 4, 8, 12: 250 mg (two 1-mL injections of 125 mg/mL Lebrikizumab).
  Weeks 6, 10, 14: Two 1-mL injections of placebo.
  Interventions: Biological: Lebrikizumab; Drug: Placebo
- 250 mg Lebrikizumab - Every 2 Weeks (Q2W) (Experimental): 250 mg Lebrikizumab administered SC once Q2W.
  Baseline and Week 2: Loading dose of 500 mg (four 1-mL SC injections of 125 mg/mL Lebrikizumab).
  Week 4, 6, 8, 10, 12, 14: 250 mg (two 1-mL SC injections of 125 mg/mL Lebrikizumab).
  Interventions: Biological: Lebrikizumab; Drug: Placebo
- Group 4 - Placebo (Placebo Comparator): Placebo administered SC once Q2W.
  Baseline and Week 2: Four 1-mL SC injections of placebo.
  Week 4, 6, 8, 10, 12, 14: Two 1-mL SC injections of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Lebrikizumab — Sterile liquid solution administered subcutaneously.
  Other Names: LY3650150; DRM06
  Arms: 125 milligrams (mg) Lebrikizumab - Every 4 Weeks (Q4W); 250 mg Lebrikizumab - Every 2 Weeks (Q2W); 250 mg Lebrikizumab - Q4W
Drug: Placebo — Solution administered subcutaneously.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of lebrikizumab compared with placebo in participants with moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older.
* Chronic AD as defined by Hanifin and Rajka (1980) that has been present for ≥1 year before the screening visit .
* Eczema Area and Severity Index (EASI) score ≥16 at the screening and the baseline visit.
* Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the screening and the baseline visit.
* ≥10% body surface area (BSA) of AD involvement at the screening and the baseline visit.

Exclusion Criteria:

* Treatment with any of the following agents within 4 weeks prior to the baseline visit:
* Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
* Phototherapy and photochemotherapy (PUVA) for AD.
* Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 1 week prior to the baseline visit.
* Treatment with:
* An investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, prior to the baseline visit.
* Dupilumab within 3 months prior to baseline visit.
* Cell-depleting biologics, including rituximab, within 6 months prior to the baseline visit.
* Other biologics within 5 half-lives (if known) or 16 weeks prior to baseline visit (whichever is longer).
* Use of prescription moisturizers within 7 days of the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (58):
- United States (58):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - University of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Stanford Medicine Outpatient Center-Medical Dermatology Clinic, Redwood City, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - UCSD Dermatology, San Diego, California
  - TCR Medical Corporation, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Total Vein and Skin, Boynton Beach, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Olympian Clinical Research, Largo, Florida
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Integrated Clinical Research, LLC, West Palm Beach, Florida
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - ActivMed Practices & Research, Inc., Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Somerset Skin Centre, Troy, Michigan
  - JDR Dermatology Research, Las Vegas, Nevada
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Schweiger Dermatology, PLLC, New York, New York
  - Icahn School of Medicine, New York, New York
  - Sadick Research Group, LLC., New York, New York
  - DermResearchCenter of New York, Inc., Stony Brook, New York
  - Piedmont Plastic Surgery and Dermatology, Charlotte, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Rivergate Dermatology Clinical Research Center, Goodlettsville, Tennessee
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Menter Dermatology Research, Dallas, Texas
  - The University of Texas Health, Houston, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Rams A, Baldasaro J, Bunod L, Delbecque L, Strzok S, Meunier J, ElMaraghy H, Sun L, Pierce E. Assessing Itch Severity: Content Validity and Psychometric Properties of a Patient-Reported Pruritus Numeric Rating Scale in Atopic Dermatitis. Adv Ther. 2024 Apr;41(4):1512-1525. doi: 10.1007/s12325-024-02802-3. Epub 2024 Feb 16. PMID 38363461
- [Derived] Guttman-Yassky E, Blauvelt A, Eichenfield LF, Paller AS, Armstrong AW, Drew J, Gopalan R, Simpson EL. Efficacy and Safety of Lebrikizumab, a High-Affinity Interleukin 13 Inhibitor, in Adults With Moderate to Severe Atopic Dermatitis: A Phase 2b Randomized Clinical Trial. JAMA Dermatol. 2020 Apr 1;156(4):411-420. doi: 10.1001/jamadermatol.2020.0079. PMID 32101256

RESULTS

PARTICIPANT FLOW:
Groups:
- 125 Milligrams (mg) Lebrikizumab - Every 4 Weeks (Q4W): 125 milligrams (mg) Lebrikizumab administered subcutaneously (SC) once every Q4W.
  Baseline: Loading dose 250 mg Lebrikizumab SC (two injections SC 1-mL of 125 mg/mL Lebrikizumab and 1-mL placebo).
  Week 2: Four 1-mL SC injections placebo.
  Weeks 4, 8, 12: 125 mg SC Lebrikizumab and 1-mL SC placebo.
  Weeks 6, 10, 14: Two 1-mL SC placebo.
- 250 mg Lebrikizumab (Q4W): 250 mg Lebrikizumab administered SC once every 4 weeks.
  Baseline: Loading dose of 500 mg (four 1-mL SC injections of 125 mg/mL Lebrikizumab).
  Week 2: Four 1-mL SC injections of placebo.
  Weeks 4, 8, 12: 250 mg (two 1-mL injections of 125 mg/mL Lebrikizumab).
  Weeks 6, 10, 14: Two 1-mL injections of placebo.
- 250 mg Lebrikizumab - Every 2 Weeks (Q2W): 250 mg Lebrikizumab administered SC once every 2 weeks.
  Baseline and Week 2: Loading dose of 500 mg (four 1-mL SC injections of 125 mg/mL Lebrikizumab).
  Week 4, 6, 8, 10, 12, 14: 250 mg (two 1-mL SC injections of 125 mg/mL Lebrikizumab).
- Placebo: Placebo administered SC once every 2 weeks.
  Baseline and Week 2: Four 1-mL SC injections of placebo.
  Week 4, 6, 8, 10, 12, 14: Two 1-mL SC injections of placebo.
Period: Overall Study
Arm/Group | 125 Milligrams (mg) Lebrikizumab - Every 4 Weeks (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab - Every 2 Weeks (Q2W) | Placebo
Started | 73 | 80 | 75 | 52
Received at Least One Dose of Study Drug | 73 | 80 | 75 | 52
Completed | 52 | 49 | 56 | 20
Not Completed | 21 | 31 | 19 | 32
Not completed — Adverse Event | 2 | 4 | 3 | 1
Not completed — Lost to Follow-up | 9 | 9 | 7 | 5
Not completed — Withdrawal by Subject | 8 | 15 | 9 | 23
Not completed — Physician Decision | 1 | 2 | 0 | 1
Not completed — Sponsor Decision | 1 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 125 mg Lebrikizumab (Q4W): 125 mg Lebrikizumab administered SC once every 4 weeks.
- 250 mg Lebrikizumab (Q4W): 250 mg Lebrikizumab administered SC once every 4 weeks.
- 250 mg Lebrikizumab (Q2W): 250 mg Lebrikizumab administered SC once every 2 weeks.
- Placebo: Placebo administered SC once every 2 weeks.
- Total: Total of all reporting groups
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo | Total
Number analyzed (Participants) | 73 | 80 | 75 | 52 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (16.54) | 40.2 (17.88) | 38.9 (17.36) | 42.2 (18.21) | 39.3 (17.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 49 | 24 | 166
  Male | 27 | 33 | 26 | 28 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 12 | 5 | 42
  Not Hispanic or Latino | 59 | 69 | 63 | 47 | 238
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 0 | 3
  Asian | 8 | 7 | 6 | 6 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 26 | 28 | 23 | 16 | 93
  White | 37 | 42 | 40 | 26 | 145
  More than one race | 1 | 2 | 5 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 80 | 75 | 52 | 280
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: units on a scale] — EASI assesses objective physician estimates of 2 dimensions of AD - disease extent & clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1)erythema, (2)edema/papulation, (3)excoriation, & (4)lichenification each on a scale of 0 to 3(0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body site (head/neck, trunk, upper limbs, & lower limbs). Half scores are allowed between severities 1, 2, & 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  units on a scale | 29.85 (13.517) | 26.15 (10.135) | 25.48 (11.206) | 28.90 (11.790) | 27.45 (11.764)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Square (LS) Means were calculated using analysis of covariance (ANCOVA) with the factor of treatment and the baseline EASI as covariate.
  Note: Missing values were imputed using Markov Chain Monte Carlo (MCMC) multiple imputation.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had Week 16 EASI data.
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Groups:
- 125 mg Lebrikizumab (Q4W): 125 mg Lebrikizumab administered SC once Q4W.
- 250 mg Lebrikizumab (Q4W): 250 mg Lebrikizumab administered SC once Q4W.
- 250 mg Lebrikizumab (Q2W): 250 mg Lebrikizumab administered SC once Q2W.
- Placebo: Placebo administered SC once Q2W.
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 73 | 80 | 75 | 52
percent change | -62.34 (37.266) | -69.21 (38.282) | -72.09 (37.229) | -41.12 (59.496)
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0165, ANCOVA
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0022, ANCOVA
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0005, ANCOVA

2. Secondary Outcome: Percentage of Participants With a 75% Improvement From Baseline in EASI (EASI75) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 73 | 80 | 75 | 52
percentage of participants | 43.3 | 56.1 | 60.6 | 24.3
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0610, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) and a Reduction ≥2 Points From Baseline to Week 16 (5-point Scale)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 73 | 80 | 75 | 52
percentage of participants | 26.6 | 33.7 | 44.6 | 15.3
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.1917, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0392, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0023, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With EASI <7 at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 73 | 80 | 75 | 52
percentage of participants | 42.2 | 61.2 | 61.8 | 29.3
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.2043, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0018, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants Achieving EASI50 at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 50% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 73 | 80 | 75 | 52
percentage of participants | 66.4 | 77.0 | 81.0 | 45.8
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0554, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0037, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants Achieving EASI90 at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 73 | 80 | 75 | 52
percentage of participants | 26.1 | 36.1 | 44.0 | 11.4
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0800, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0062, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percent Change From Baseline in the Sleep Loss Scale Score
Description: The Sleep Loss Scale is used by the participants to report the impact of itching on their sleep every night. Participants responded to the question to what extent did your itching interfere with your sleep last night. The scale ranged from 0 to 4, with 0 (not at all) to 4 (unable to sleep at all). Higher scores indicated a greater impact and worse outcome. Assessments were recorded daily by the participant using an electronic diary.
  Least Squares (LS) Means were calculated using ANCOVA with the factor of treatment and the baseline sleep-loss scale as covariates.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had Week 16 Sleep Loss Scale score.
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 38 | 33 | 38 | 14
percent change | -48.68 (50.692) | -53.03 (50.662) | -64.69 (50.692) | -20.24 (51.066)
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0773, ANCOVA
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0459, ANCOVA
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0062, ANCOVA

8. Secondary Outcome: Percent Change From Baseline in Pruritus Numeric Rating Score (NRS)
Description: The Pruritus NRS is an 11-point scale used by participants to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating worst itch imaginable. Pruritus assessments were recorded daily by the participant using an electronic diary.
  LS Means were calculated using ANCOVA with the factor of treatments and the baseline pruritus NRS as covariates.
Time Frame: Baseline, Week 16
Population: All randomized participants who received least one dose of study drug and had Week 16 Pruritus NRS score.
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 55 | 56 | 50 | 22
percent change | -35.94 (55.553) | -49.60 (55.555) | -60.63 (55.564) | 4.26 (55.610)
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0047, ANCOVA
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

9. Secondary Outcome: Percentage of Participants With Pruritus NRS Change of ≥3 at Week 16
Description: The Pruritus NRS is an 11-point scale used by participants to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating worst itch imaginable. Assessments were recorded daily by the participant using an electronic diary.
  The percentage of participants who are dichotomized to success (pruritus NRS greater than or equal to 3-point improvement) at Week 16 will be analyzed using a Cochran-Mantel-Haenszel (CMH) test.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug and had a >=3 point improvement from Baseline in Week 16 Pruritus NRS score.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 55 | 57 | 50 | 22
percentage of participants | 50.9 | 64.9 | 76.0 | 45.5
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.6674, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.1166, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0119, Cochran-Mantel-Haenszel

10. Secondary Outcome: Percentage of Participants With Pruritus NRS Change of ≥4 From Baseline to Week 16
Description: The Pruritus NRS is an 11-point scale used by participants to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating worst itch imaginable. Assessments were recorded daily by the participant using an electronic diary.
  The percentage of participants who are dichotomized to success (pruritus NRS greater than or equal to 4-point improvement) at Week 16 will be analyzed using a Cochran-Mantel-Haenszel (CMH) test.
Time Frame: Week 16
Population: All randomized participants who received at least one dose of study drug and had a >=4 point improvement from Baseline in Week 16 Pruritus NRS score.
Measure: Number; unit: percentage of participants
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 55 | 57 | 50 | 22
percentage of participants | 41.8 | 47.4 | 70.0 | 27.3
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.2371, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.1067, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel

11. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Involved With Atopic Dermatitis (AD)
Description: The body surface area (BSA) affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). Percent of BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had Week 16 BSA data.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 59 | 62 | 59 | 24
percentage of BSA | -19.6 (19.08) | -24.9 (20.08) | -24.3 (21.00) | -17.4 (20.56)
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.4631, ANCOVA
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0368, ANCOVA
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0232, ANCOVA

12. Secondary Outcome: Change From Baseline in Atopic Dermatitis Impact Questionnaire (ADIQ) Score
Description: The ADIQ is a 17-item questionnaire used to assess the participant's AD-specific health-related quality of life. Each item is rated on a 5-point scale from 0 to 4, with higher numbers indicating greater burden. The questionnaire assesses AD's impact on emotions, energy, activities of daily living, and social activities. The ADIQ has a recall specification of 7 days. Assessments were recorded by the participant using an electronic diary and transferred to the clinical database.The ADIQ score is calculated by summing the score of each of the 14 questions resulting in a maximum of 56 and a minimum of 0, with higher scores indicating greater burden.
Time Frame: Baseline, Week 16
Population: All randomized participants who received at least one dose of study drug and had evaluable Week 16 ADIQ data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
Number analyzed (Participants) | 38 | 33 | 35 | 17
score on a scale | -14.2 (12.74) | -18.8 (12.03) | -18.6 (12.63) | -11.0 (13.96)
Statistical Analysis 1: Comparison: 125 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.4729, ANCOVA
Statistical Analysis 2: Comparison: 250 mg Lebrikizumab (Q4W) vs Placebo; Test type: Superiority; p = 0.0282, ANCOVA
Statistical Analysis 3: Comparison: 250 mg Lebrikizumab (Q2W) vs Placebo; Test type: Superiority; p = 0.0506, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline up to 271 days
Description: All participant who received at least one dose of study drug.
  Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 125 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q4W) | 250 mg Lebrikizumab (Q2W) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/80 | 0/75 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/80 | 2/75 | 2/52
Other Adverse Events (participants affected / at risk) | 41/73 | 39/80 | 45/75 | 24/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 125 mg Lebrikizumab (Q4W) (N=73) | 250 mg Lebrikizumab (Q4W) (N=80) | 250 mg Lebrikizumab (Q2W) (N=75) | Placebo (N=52)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 125 mg Lebrikizumab (Q4W) (N=73) | 250 mg Lebrikizumab (Q4W) (N=80) | 250 mg Lebrikizumab (Q2W) (N=75) | Placebo (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Injection site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 3 (6) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (8) | 4 (20) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2/46 (3) | 0/47 (0) | 0/49 (0) | 0/24 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0/46 (0) | 1/47 (1) | 0/49 (0) | 0/24 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (5) | 2 (3) | 9 (11) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 9 (10) | 2 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Viral tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/46 (2) | 0/47 (0) | 0/49 (0) | 0/24 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/46 (0) | 1/47 (1) | 1/49 (1) | 0/24 (0)
Vulvovaginitis gonococcal (Infections and infestations) | 0/46 (0) | 0/47 (0) | 0/49 (0) | 1/24 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Auditory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/46 (0) | 0/47 (0) | 0/49 (0) | 1/24 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0/46 (0) | 0/47 (0) | 1/49 (1) | 0/24 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/46 (0) | 0/47 (0) | 1/49 (1) | 0/24 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fragility (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT03443024/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03443024/SAP_001.pdf